CLINICAL TRIAL: NCT07228572
Title: Clinical Evaluation of Resin Nanoceramic Crown Restoration for Posterior Teeth Fabricated by Three-Dimensional (3D) Printing: Short-Term Clinical Study
Brief Title: Clinical Evaluation of Three-Dimensional (3D) Printing Resin Nanoceramic Crown Restoration.
Status: Active, not recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Ege University (Other)
Collaborators: Ege University Scientific Research Projects Coordination (Unknown)
Responsible Party: Principal Investigator, ola salama, research assistant, Ege University
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Other
Other Study IDs: EGE-DHF-OS-01
Record Dates: First submitted 2025-11-13; First posted 2025-11-14 (Actual); Last update posted 2025-11-14 (Actual); Status verified 2025-11

CONDITIONS: 3d Printing Ceramic Restoration; Nanoceramic Crown Restoration for Posterior Teeth
Keywords: nanoceramic crown; 3d printed

STUDY DESIGN:
Intervention Model Description: case - control study
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- nanoceramic crown restorations ; clinical evolution (Experimental): the crown preparation for the tooth of each patient included in the study will be perfomered using preparation bur set under water cooling with a rotary handpiece. then digital impression of the prepared teeth will be obtained using an intra-oral scanner to facilitate the design of crown restorations. following their design and fabrication, the 3d printed nanoceramic crown restorations will be adhesively cemented to the teeth after verifying their fit.
  Interventions: Other: 3D printing hybrid ceramic crown restorations

INTERVENTIONS:
Other: 3D printing hybrid ceramic crown restorations — crown restorations fabricated with 3D printing nanoceramic will be applied to 60 patients. following the 6 and 12 month follow-ups, the collected data will be analyzed according to clinical evaluation criteria.

SUMMARY:
This study aims to evaluate the function and aesthetics of ceramic-filled hybrid resin permanent crowns produced by 3D printing method in posterior teeth according to Revised FDI criteria.

At the Department of Prosthodontics, Faculty of Dentistry, Ege University, 60 patients who present for single-tooth crown restoration in the posterior region of either the maxilla or mandible and who meet the inclusion criteria will receive a total of 60 permanent crown restorations. Following tooth preparation, the restorations will be fabricated using a three-dimensional (3D) printing technique with a ceramic-filled hybrid resin material (VarseoSmile TriniQ, Bego, Bremen, Germany).

The effects of restorations on clinical success will be evaluated according to demographic data (age, gender, etc.) and modified USPHS and Revised FDI criteria, and statistical analysis will be applied to the recorded data. Follow-up visits are scheduled at 0: baseline, 6, and 12 months.

DETAILED DESCRIPTION:
The study will be conducted between June 2025 and June 2026. Tooth preparation will be performed following clinical and radiographic examinations. The study schedule will be explained in detail to all patients included in the study.

According to the power analysis performed (G*Power Ver. 3.0.10), at a significance level of p= 0.05, the inclusion of at least 16 patients was determined to be necessary to achieve a statistical power of at least 80%. To further increase the power of the study, it was planned to include 60 patients who meet the inclusion criteria.

Eligible patients will be provided with detailed and comprehensible information regarding the content of the study. Subsequently, the informed consent form will be presented and read, and any questions from the patient will be addressed. If the patient agrees to participate in the study, the form will be signed.

Prosthetic treatment phase:

In the clinics of the Department of Prosthodontics, Faculty of Dentistry, Ege University, following completion of tooth preparation, crown restorations will be fabricated from a ceramic-filled permanent hybrid resin material (VarseoSmile TriniQ, Bego, Bremen, Germany) using a 3D printing technique, based on intraoral optical scans obtained with an intraoral scanner (iTero 5D Element Plus, Align Technology, USA). The restorations will be cemented with a self-adhesive resin cement Panavia V5 Standard Kit (Kuraray Noritake, Osaka, Japan). Occlusion will be checked, and patients will be provided with routine oral hygiene instructions.

Clinical and radiographic evaluations of 3D-printed crowns will be performed at 6 and 12 months. Data will be recorded according to the revised FDI criteria and modified united states public health service USPHS criteria.

At each follow-up visit, patients' teeth will be scanned using intraoral scanner (iTero 5D Element Plus, Align Technology, USA). The STL files of scans will be superimposed using Geomagic software, and the wear will be evaluated.

ELIGIBILITY:
Inclusion Criteria:

* Individuals between 18 and 65 years of age, Patients requiring a single crown restoration in the posterior region of the maxilla or mandible, Absence of active periodontal disease, Presence of an opposing tooth (natural or restored), Presence of adjacent teeth (mesial and distal), Vital or endodontically treated (devital) teeth without periapical lesions, Patients who agree to comply with the study conditions will be included in the study.

Exclusion Criteria:

* Suspected or confirmed pregnancy, or patients in the breastfeeding period, Teeth requiring coverage that are intended to serve as abutments for fixed partial dentures, Vital or endodontically treated (devital) teeth with periapical lesions, Absence of an opposing tooth or presence of an opposing tooth restored with a crown, Absence of adjacent teeth (mesial or distal), Individuals with temporomandibular joint disorders (TMDs), patients who do not consent to the study conditions will be excluded from the study.

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 60 (Estimated)
Dates: Start 2025-06-26 (Actual); Primary Completion 2026-06 (Estimated); Study Completion 2026-09 (Estimated)

PRIMARY OUTCOMES:
Revised FDI criteria for evaluating direct and indirect dental restorations | one year
  In 2007, an international workgroup published new FDI criteria to evaluate the quality of direct and indirect restorations; an update with clinical cases was published in 2010. Then, these criteria are revised in 2022. This diagnostic system classified aesthetic, functional, and biological properties and covers various types of failures by using 16 different categories with five grades for each criterion. In detail, scores 1 to 3 indicated clinically acceptable restorations, and scores 4 and 5 summarized clinically unacceptable situations indicating repair (score 4) or replacement (score 5).
Modified united states public health service (USPHS) criteria | one year
  The clinical performance of crown restorations are evaluated by using USPHS criteria. Parameters such as color match, anatomic form, marginal integrity, surface roughness, retention and post-operative sensitivity are assessed. Each parameter is scored using Alpha, Bravo and Charlie ratings. Alpha indicates to optimal clinical performance, Bravo rating is for an acceptable level and Charlie rating represents the need for restoration repair or replacement.

CONTACTS AND LOCATIONS:
Locations (1):
- Ege University, Faculty of Dentistry, Department of Prosthodontics, Izmir, İzmir, Turkey (Türkiye)